CLINICAL TRIAL: NCT03781050
Title: Efficacy of Rapamycin (Sirolimus) in the Treatment of Peutz-Jeghers Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-1607
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Peutz-Jeghers Syndrome
Keywords: Peutz-Jeghers Syndrome (PJS); Rapamycin (sirolimus); Mammalian target of rapamycin (mTOR) inhibitor; Treatment
MeSH Terms: conditions — Peutz-Jeghers Syndrome; Hereditary Sensory and Autonomic Neuropathies | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapamycin (Experimental): For children: rapamycin, 1 mg per square meter of body surface area a day, orally, for at least 6 months
  For adults: rapamycin, 2 mg a day, orally, for at least 6 months
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — For children: rapamycin, 1 mg per square meter of body surface area a day, orally, for at least 6 months
  For adults: rapamycin, 2 mg a day, orally, for at least 6 months
  Other Names: Sirolimus

SUMMARY:
A prospective non-randomized open label single arm clinical trial to examine the efficacy and safety of sirolimus in patients with Peutz-Jeghers Syndrome.

DETAILED DESCRIPTION:
PJS (Peutz-Jeghers Syndrome) is mostly caused by mutations in Lkb1 gene, which leads to an increased activity of mTOR pathway, thus making mTOR inhibitor (sirolimus) a promising candidate in treatment and prevention of PJS. The efficacy of sirolimus (rapamycin) on PJS has been demonstrated in mouse model, but no clinical trials have been reported. Our study was designed as a prospective non-randomized open label single arm clinical trial to examine its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with PJS.
* Patients have gastrointestinal polyps related syndromes, including abdominal pain, abdominal distension, gastrointestinal bleeding, etc, with imageological examination suggesting intestinal obstruction or intussusception; or whose symptoms recur after previous digestive endoscopic treatment and surgery; or who are inappropriate or unwilling to accept the above treatment again and wish to receive pharmacotherapy.
* Conventional treatment didn't work well in patients combined with PJS-related tumors.
* Physical condition (ECGO): 0~3
* Organ function is good and biochemical indices meet the following conditions:

  * AST≤2.5×upper limit of normal value (ULN),
  * ALT≤2.5×upper limit of normal value (ULN),
  * Serum total bilirubin (TSB)≤1.5×upper limit of normal value (ULN),
  * Creatinine≤1.5×upper limit of normal value (ULN).
* No other medications have been received for intestinal polyps within 3 months prior to the clinical trial.
* Patients participate in the trial voluntarily and have signed the informed consent by the participant or his/her legal guardian.

Exclusion Criteria:

* Patients underwent a surgery within 2 weeks.
* Patients may need emergency surgery in the near future.
* Patients are allergic to any ingredient of rapamycin.
* Patients suffer from a disease requiring immediate blood transfusion.
* Patients suffer from any disease or condition that may impact implementation of the study or interpretation of the results. This type of diseases includes:

  * Known severe blood coagulation disorders
  * Known anemia that is not caused by intestinal polyps
  * Known hemoglobinopathy
  * Other gastrointestinal infectious diseases
  * Serious heart, liver, kidney and other concomitant diseases that may endanger lives
* Patients are in pregnancy and lactation.
* Alcohol or drug (such as aperient) abuse
* Patients took part in another clinical trial that may influence this study.
* The researchers believe that there are other unfavorable reasons for the patient to become a subject.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09-16 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Total load of PJS-related intestinal polyps Total load of PJS-related intestinal polyps Total load of PJS-related intestinal polyps | The time from start of therapy to 1 year
  Lesion load (cm2) = A+B. A = sum of the product of maximum diameter and maximum height of the largest 3 lesions shown by abdomen and pelvis MRI or small bowel CT reconstruction (in cm2). B = sum of the product of maximum diameter and maximum height of the largest 3 lesions shown by digestive endoscope (in cm2). Remarks: 1. If it is impossible to evaluate 3 or more lesions, results of the actual number of lesions should be taken as valid; 2. Lesions evaluated should be correspondent before and after treatment. If the lesion is difficult to assess after treatment, it should be ruled out from the assessment.

SECONDARY OUTCOMES:
Concentration of hemoglobin in blood | The time from start of therapy to 1 year
  The value indicates the amount of gastrointestinal bleeding.
Concentration of albumin in blood | The time from start of therapy to 1 year
  The value indicates the status of nutrition.
Concentration of hsCRP in blood | The time from start of therapy to 1 year
  The value indicates the level of inflammation.
Visual analogue score (VAS) | The time from start of therapy to 1 year
  The value indicates the level of pain.
Dermatology life quality index (DLQI) | The time from start of therapy to 1 year
  The value indicates the status of hyperpigmented macules on the lips and oral mucosa.
Adverse events | The time from start of therapy to 1 year
  To evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Jiaolin Zhou, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, China/Beijing, China

REFERENCES:
- [Background] Chen HY, Jin XW, Li BR, Zhu M, Li J, Mao GP, Zhang YF, Ning SB. Cancer risk in patients with Peutz-Jeghers syndrome: A retrospective cohort study of 336 cases. Tumour Biol. 2017 Jun;39(6):1010428317705131. doi: 10.1177/1010428317705131. PMID 28653895
- [Background] Shaw RJ, Bardeesy N, Manning BD, Lopez L, Kosmatka M, DePinho RA, Cantley LC. The LKB1 tumor suppressor negatively regulates mTOR signaling. Cancer Cell. 2004 Jul;6(1):91-9. doi: 10.1016/j.ccr.2004.06.007. PMID 15261145
- [Background] Jenne DE, Reimann H, Nezu J, Friedel W, Loff S, Jeschke R, Muller O, Back W, Zimmer M. Peutz-Jeghers syndrome is caused by mutations in a novel serine threonine kinase. Nat Genet. 1998 Jan;18(1):38-43. doi: 10.1038/ng0198-38. PMID 9425897
- [Background] Wei C, Amos CI, Zhang N, Zhu J, Wang X, Frazier ML. Chemopreventive efficacy of rapamycin on Peutz-Jeghers syndrome in a mouse model. Cancer Lett. 2009 May 18;277(2):149-54. doi: 10.1016/j.canlet.2008.11.036. Epub 2009 Jan 14. PMID 19147279
- [Background] Robinson J, Lai C, Martin A, Nye E, Tomlinson I, Silver A. Oral rapamycin reduces tumour burden and vascularization in Lkb1(+/-) mice. J Pathol. 2009 Sep;219(1):35-40. doi: 10.1002/path.2562. PMID 19434632

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03781050/Prot_SAP_000.pdf